CLINICAL TRIAL: NCT03420131
Title: DETErmining the funCTional Significance of Intermediate Stenoses in isCHEMIc heArt Disease (DETECT ISCHEMIA): Diagnostic Agreement of iFR and QFR.
Brief Title: Diagnostic Agreement of iFR and QFR.
Acronym: DETECTISCHEMIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Contilia Clinical Research Institute (Other)
Responsible Party: Principal Investigator, Christoph Jensen, MD Associate Prof., Christoph Jensen, MD, Associate Professor of medicine, Contilia Clinical Research Institute
Other Study IDs: U1111-1199-4364
Record Dates: First submitted 2018-01-27; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Fractional Flow Reserve, Myocardial; Coronary Artery Disease
Keywords: instantaneous Flow Ratio; Quantitative Flow Ratio; Fractional Flow Reserve
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FFR-iFR-QFR group
  Interventions: Diagnostic Test: QFR and iFR

INTERVENTIONS:
Diagnostic Test: QFR and iFR — iFR® (CE-Marked) is a pressure-derived, hyperemia-free index for the assessment of coronary stenosis relevance. This option consists of an FFR-iFR® specific patient interface module (PIM-FFR) which can be connected to the Volcano system - VOLCANO s5 or s5i™ platform equipped with iFR® option.
  QFR® (CE-Marked) is an angio-based FFR estimation using the analytical Software QAngio XA 3D from Medis medical imaging B.V., The Netherland

SUMMARY:
A Prospective, observational, single center diagnostic study to investigate the the diagnostic agreement between QFR and the pressure wire-based iFR in a real world setting.

DETAILED DESCRIPTION:
During coronary angiography, intermediate stenoses can not be adequately assessed by visual assessment alone. It is necessary to evaluate the functional significance to guide their treatment.

Fractional Flow Reserve (FFR) is the current gold standard for determining this functional significance but its adoption in clinical practice remains low. The instantaneous wave-free ratio (iFR) is an alternative way to determine the flow-limiting characteristics of a coronary stenosis with a pressure wire but without the need to induce hyperemia. Large randomised trials have confirmed the non-inferiority of iFR in respect to FFR in terms of outcome.

Quantitative Flow Ratio (QFR) is another new method for evaluating the functional significance of coronary stenosis It is a software-based analysis of conventional angiographic images to estimate the pressure drop caused by a coronary stenosis. The diagnostic agreement with FFR seemed promising in the FAVOR Pilot Study and a larger trial is enrolling for confirmation.

A stepwise approach of QFR and iFR could make the functional assessment of intermediate stenoses more practical and cost-effective. However before being used as a combination in daily practice, QFR has to be validated in respect to iFR.

The primary objective of the trial is to investigate the diagnostic agreement between QFR and the pressure wire-based iFR in a real world setting

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 with symptoms of myocardial ischemia and angina or angina equivalent (chest pain, abnormal stress testing, abnormal noninvasive testing)
* Patients witch semi recent (>3 days) acute coronary syndromes can be included but only for the non-culprit vessels and outside of primary intervention during acute myocardial infarction.
* Willing to participate and able to understand, read and sign the informed consent document before the planned procedure
* Eligible for coronary angiography and/or percutaneous coronary intervention
* Coronary artery disease with at least 1 or more visually assessed de novo coronary stenosis (30-90% diameter stenosis) in native major epicardial vessel or its branches by coronary angiogram.

Exclusion criteria:

* Contraindication to adenosine administration
* Previous Coronary Artery Bypass surgery with patent grafts to the interrogated vessel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that undergo angiography because of symptoms of myocardial ischemia and angina or angina equivalent (chest pain, abnormal stress testing or abnormal noninvasive testing) and in whom hemodynamic evaluation of an intermediate stenosis is indicated should be screened and considered for participation in the trial
  The trial design is set up to be representative for the patient population that under current guidelines should be evaluated with FFR. Therefore the exclusion criteria are limited to the contraindications for adenosine and previous CABG which would not allow accurate evaluation by FFR and QFR respectively.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-07-18 (Actual); Primary Completion 2018-07-28 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of QFR in comparison to iFR | 1 hour
  reported as sensitivity, specificity, positive and negative likelihood ratio of QFR according to iFR
QFR- iFR diagnostic grey zone calculation. | 1 hour
  QFR limits for achieving 95% sensitivity and specificity in comparison to iFR

SECONDARY OUTCOMES:
Diagnostic performance of QFR in comparison to FFR | 1 hour
  reported as sensitivity, specificity, positive and negative likelihood ratio of QFR according to FFR
QFR- FFR diagnostic grey zone calculation. | 1 hour
  QFR limits for achieving 95% sensitivity and specificity in comparison to FFR
Diagnostic performance of iFR in comparison to FFR | 1 hour
  reported as sensitivity, specificity, positive and negative likelihood ratio of iFR according to FFR
iFR- FFR diagnostic grey zone calculation. | 1 hour
  iFR limits for achieving 95% sensitivity and specificity in comparison to FFR
effect of 3D QCA characteristics on QFR-iFR-FFR disagreement. | 1 hour
  Influence of minimum luminal area (MLA), percentage area stenosis, lesion length, and minimum luminal diameter (MLD) and percentage diameter stenosis in the prediction of QFR-iFR-FFR disagreement.
Effect of lesion location on QFR-iFR-FFR disagreement. | 1 hour
  Evaluation of lesion location in the prediction of QFR-iFR-FFR disagreement.
Effect of p20-DAC2 score in proximal and mid-LAD stenosis on QFR-iFR-FFR disagreement. | 1 hour
  Evaluation of p20-DAC2 score in proximal and mid-LAD stenosis in in the prediction of QFR-iFR-FFR disagreement.

OTHER OUTCOMES:
Cost analysis | 1 hour
  Cost savings of removing the need for Adenosine by using iFR. Evaluation of costs by excess/reduced need for stenting when iFR and FFR disagree

CONTACTS AND LOCATIONS:
Overall Officials: Christoph j Jensen, MD, Principal Investigator — contilia heart and vascular center
Locations (1):
- Contilia heart and vascular center, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided